CLINICAL TRIAL: NCT03915600
Title: Evaluation of the Citotoxicity and Clicemic Control of Subject With Metabolic Syndrome Managed With Conventional Nutritional Tratment More Quinoa, Flaxseed or Borh Versus Conventional Nutrition
Brief Title: Efect of Quinoa and Flaxseed in Cititoxicity and Glicemic Control in Metabolic Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Ana Lilia Fletes Rayas, PROFESSOR ASSOCIATE TYPE A, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 235/15
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-04

CONDITIONS: Metabolic Syndrome; Nutritional and Metabolic Diseases
Keywords: Metabolic Syndrome; Micronuceli; Quinoa; Flaxseed; Diet
MeSH Terms: conditions — Metabolic Syndrome; Nutritional and Metabolic Diseases | interventions — chenopodin protein, Chenopodium quinoa; Linseed Oil

STUDY DESIGN:
Intervention Model Description: An open clinical trial with randomization plus control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Quinoa (Experimental): Personalized diet added with quinoa
  Interventions: Other: Quinoa
- Flaxseed (Experimental): Personalized diet added with Flaxseed
  Interventions: Other: Flaxseed
- Quinoa and Flaxseed (Experimental): Personalized diet added with quinoa and flaxseed
  Interventions: Other: Quinoa and Flaxseed
- Normal diet (No Intervention): Personalized diet without dietary supplement

INTERVENTIONS:
Other: Quinoa — Personalized diet added with quinoa
  Arms: Quinoa
Other: Flaxseed — personalized diet added with flaxseed
  Arms: Flaxseed
Other: Quinoa and Flaxseed — personalized diet added with quinoa and flaxseed
  Arms: Quinoa and Flaxseed

SUMMARY:
The Metabolic Syndrome (MS) is a set of anthropometric alterations and chronic-degenerative diseases, such as obesity, diabetes mellitus and arterial hypertension. Each one of the diseases and physiological alterations represents a risk factor that conditions in the medium or long term another incapacitating or limiting disease that reduces the quality of life of an individual.

Our country has a growing burden of morbidity and mortality due to diseases chronic-degenerative caused, for the most part, to the unhealthy lifestyle produced by multiple factors, such as social, economic, behavioral, environmental, among others. For this reason, it is important to plan, design and implement strategies that reduce, mitigate or control this public health problem in the population. The purpose of this study is to perform a nutritional intervention that includes food such as quinoa, flaxseed or both in subjects with metabolic syndrome and follow them up for six months. The impact of this intervention will be carried out through the measurement of cytotoxicity and glycemic control, this is with the micronucleus count and the estimation of glycosylated hemoglobin (Hba1c).

This document will explain in detail what is intended to be done by presenting the following sections:

In the approach of the problem and the justification, the metabolic syndrome will be described, its impact on the Mexican population, the interest and relevance of this research project.

In the background will be detailed what has been said and done in the different studies scientists regarding the consumption of quinoa and flaxseed. Methodology defines the strategy, conditions, clinical criteria, material and epidemiological and statistical methods for the management of subjects and information.

DETAILED DESCRIPTION:
The "strong pulse disease" was treated by acupuncture, phlebotomy and leeches from 2600 to c. Modern history began when in 1628 William Harvey described the circulatory system and in 1733 stephen hales made the first blood pressure measurement. In 1896 was recognized as a clinical entity, thanks to the invention of the sphygmomanometer by Riva-rocci and in 1913 janeway coined the term "hypertensive vascular disease". The metabolic syndrome was described since 1988 as syndrome x, with the intention of showing how the cardiovascular risk factors are grouped together: obesity, hyperglycemia, dyslipidemia and arterial hypertension. Earlier, in 1920, Kylin had described that diabetes, high blood pressure and gout were associated, but not related to cardiovascular disease. Syndrome x was later called insulin resistance syndrome and, finally, metabolic syndrome or cardiometabolic syndrome. By 1999, the world health organization reported what would be the first diagnostic criteria for the metabolic syndrome. Soon they were reason for criticism because they were considered impractical, because it was necessary to diagnose insulin resistance and microalbuminuria. From then to date numerous criteria have been reported, perhaps the most used to date, in adults they are the

3.- NCEP-ATPIII (from the third treatment panel of adults of the national cholesterol education program of the United States). The main trigger of this conglomerate of atherogenic, prothrombotic, proinflammatory and metabolic factors is obesity, in our country, the prevalence of overweight and obesity in adults increased from 62 to 70% in just five years. In the last century, in Mexico the energy density of the diet was increased by almost 24% (26% more carbohydrates and 36% more fat) and physical activity has been reduced In Mexico, the prevalence of metabolic syndrome in children and adolescents is 20% and is strongly linked to overweight and childhood obesity.

Mexicans are world leaders in obesity, since one in three Mexicans is overweight due to poor diet. In February 2012, the organization for cooperation and economic development (OECD) reported that Mexico was the second most overweight or obese country on a list that includes 40 nations, adding that three out of seven Mexicans have a waistline bigger than they should be. Chronic degenerative diseases have displaced infectious diseases as the main causes of mortality in Mexico. In 2011, 70 of every 100.00 people died from this disease in the country.

In Mexico, aguilar-salinas reported an age-adjusted prevalence of 13.6% with the criterion of the world health organization and 26.6% with the ncep-atpiii criterion in people between 20 and 69 years old, from the ensa survey. -2000; while González-Villalpando in the Diabetes Study of Mexico City reported prevalences of 39.9 and 59.9% for men and women, respectively, based on the criteria of the Ncep-ATP III.

In Mexico, diabetes is the leading cause of blindness acquired in the productive age; as well it is the first cause of non-traumatic amputations of the lower limbs and of chronic renal failure. Short and long-term complications require medical attention and specialized treatments, which means that your care entails overwhelmingly high costs. The Binomial insulin resistance/hyperinsulinemia are associated with a significant increase in cardiovascular morbidity and mortality expressed as atherosclerosis, acute cerebral, cardiac or peripheral ischemic syndromes, as well as other pathologies, which due to their coexistence and physiopathological co-responsibility has been called metabolic syndrome.

In 2011 Mexico ranked ninth in the world in the prevalence of diabetes and the projections indicate that by the year 2025, the country will occupy the sixth or seventh place. Diabetes mellitus is defined as a chronic disease that involves a heterogeneous group of disorders that alter the production and use of insulin by the body. The most frequent modality is type 2, which occurs in adults, although it is increasingly appearing in young people and children. When there are sustained increases in blood glucose, decompensation and complications occur.

Therefore, although diabetes is an endocrine disease in its origin, its main manifestations are those of a metabolic disease. On average, men with diabetes die at a younger age than women (67 versus 70 years respectively) and only 20% of men who have developed this condition live more than 75 years, compared to 26% in the case of women. In a study conducted in Mexico by Arredondo and Icazaen 2011, the direct costs of care for the disease were calculated in all institutions of the health sector and private insurance, which amounted to $ 343,226,541 m.n. in terms of indirect costs, they were estimated around $ 778,427, 475 m.n. It is important to emphasize that for every 100 pesos spent on diabetes in Mexico, approximately 51 pesos comes from households / family income, which represents a social burden of very high impact. Regarding direct costs, of every 100 pesos spent on diabetes in Mexico, 52 are spent on 10% of the population, 33 on 48% (insured) of the population and 15 pesos on the remaining 42% of the population. population (uninsured), so, in terms of allocation and flow of economic resources, the problems of inequity and access to health are evident depending on the group to which the patients and their families belong.

During the last decades, mortality due to cardiovascular diseases has increased, until it has become the leading cause of death in the United Mexican States.

Atherosclerosis is among the main causes for the development of these diseases. Atherosclerosis plays a central role in three of the first five causes of death in Mexico. Atherosclerosis is a multifactorial process caused by risk factors that damage the endothelium chronically. Among which are the age, inheritance, smoking, sedentary lifestyle, unhealthy diet, elevation of systemic blood pressure, overweight and obesity, elevation of glucose levels as well as inadequate serum lipid levels. Dyslipidemias are one of the main modifiable factors of cardiovascular risk. The scrutiny and treatment of dyslipidemias is cost-effective in the entire population over 20 years of age. In addition, dyslipidemias and arterial hypertension are frequently associated and have a synergistic effect on cardiovascular risk. The results of the national health and nutrition survey 2006, show that overweight and obesity are problems that affect 70% of the population between 30 and 65 years of age, the prevalence of diabetes by previous medical diagnosis and of finding of the survey in adults at national level was 14.42%, the prevalence of hypertension was 30.8%. The general prevalence of hypercholesterolemia was 26.5%, with 28.8% in women and 22.7% in men.

Situation of overweight and obesity. A reflection of national nutrition surveys in Mexico. In 2006, according to the results of the ENSANUT, one in three men or women Teenagers are overweight or obese. This represents around 5,757, 400 adolescents in the country. The prevalence of overweight and obesity of women aged 12 to 19 in 2006 was compared with that of 1999, using the criteria proposed by the IOTF. There is a modest increase in overweight from 21.6 to 23.3 (7.8%) and a small absolute increase, but high in relative terms, in obesity: from 6.9 to 9.2 (33.3%). The prevalence of overweight, but especially that of obesity, tended to increase with age up to 60 years; in ages of 60, 70 and over 80 years, the trend of both conditions decreased, both in men and women.

Quinoa The quinoa (chenopodium quinoa willd., Amaranthaceae), an ancient crop of the mountains of the Andes of South America, has quickly gained popularity as a food functional and nutraceutical. Due to its properties the organization of agriculture and food nations launched the international year of quinoa in 2013 to promote global production, consumption, preservation and development of the biodiversity of this crop. It has more than three thousand varieties or ecotypes, both cultivated and wild, that can be summarized in five basic categories according to the altitudinal gradient: ecotypes of the sea level, the altiplano, the inter-Andean valleys, the salt flats and the yungas. It is a grain that has outstanding intrinsic characteristics, such as: its wide genetic variability, whose genetic pool is extraordinarily strategic to develop superior varieties (precocity, color and grain size, resistance to biotic and abiotic factors, the yield of grain and by-products). It has a protein of high biological value for its high content of lysine and its balance of essential amino acids, is comparable to animal protein. It is widely used, both in human and animal feed, using the leaves and tender stems as leafy vegetables, until the phase of the beginning of the panning, then the tender panicles are consumed in replacement of inflorescence vegetables, and the ripe grain, directly or processed.

Minerals: magnesium, zinc, iron and potassium. Unfortunately, quinoa contains phytic acid that can break down these minerals and reduce their absorption digestive touch.

Fitoecdisteroides: containing a wide range of therapeutic effects in mammals, including anabolic, increasing in performance, anti osteoporotic, and wound healing property.

flavonoids: these are natural antioxidants of plants, which provide multiple health benefits. Two of the best known flavonoids are kaempferol and quercetin, which is found in large quantities in quinoa. The amount of quercetin present in quinoa is higher than high superfoods in quercetin such as blueberries. These molecules have been shown to have anti-inflammatory, antiviral, anti-depressant, anti-carcinogenic properties, although until now only in animal studies. There is a lack of studies in humans.

Antioxidants This implies that you have several substances that help you get rid of free radicals, which are responsible for aging and cardiovascular diseases and cancer. In a comparison study between 10 foods it was found that quinoa had the highest amount of antioxidants.

Flaxseed Flaxseed corresponds to the flax seed (linum usitatissimum L.) and has been traditionally used as an oilseed. In recent decades there has been great interest in it due to the recognition that some of its components offer potential benefits for the maintenance of health and the prevention of some chronic noncommunicable diseases. Among these compounds with biological activity include alpha-linolenic acid, lignans and dietary fiber. Flax seed contains various compounds that can offer health benefits such as reduced risk of developing cardiovascular diseases, mitigating the effects of diabetes, kidney diseases, obesity, cancer of the colon and rectum, reduction of serum cholesterol level and promotion of intestinal evacuation.

Functional foods are foods that resemble traditional ones, but that differ from them in that they offer benefits beyond their nutritional and energetic value, in the promotion and prevention of some chronic diseases such as cardiovascular diseases, cancer, disorders of the autoimmune system , diabetes, arthritis and arrhythmia.

In recent years, the use of linseed (Linum usitatissimum L.) has been promoted as a functional food for its health benefits, mainly attributable to its content of omega-3 fatty acids, lignans, and dietary fiber (Ostojich, 2012). Due to its exclusive nutrient profile and its potential to affect the risk and development of cardiovascular diseases and some cancers, especially those dependent on hormones such as breast and prostate, it was also found effective in reducing the levels of hemoglobin A1c and cholesterol in individuals with cholesterol and high blood sugar.

Cytotoxicity and micronuclei in oral mucosa. The micronuclei are complete chromosomes or fragments of these that remain outside the cell nucleus during mitosis, the study of these can give information about the cytotoxicity, as well as environmental effects, as occupational. Cytotoxicity is mediated by intrinsic and environmental elements in which the individual is exposed, such is the case of the increased presence of micronuclei in metabolic syndrome as in diabetic patients, in the literature it has been reported that the consumption of foods rich in antioxidants could decrease the number of micronuclei.

The oral cavity has been described as a tissue in which changes associated with illness can be observed, as well as exposure to tobacco, alcoholism, or other harmful substances, as well as various entities where there are deficiencies of vitamins and antioxidants, can also assess side effects of exposure to chemotherapy or radiotherapy because the latter can affect the proliferative capacity of epithelial cells and even of the oropharyngeal tissue that can reach ulcers due to thinning.

The characteristics that can be observed in the micronucleus test are the following:

Normal cells: the nucleus of these is uniformly dyed, it can be round or oval. These cells are considered as totally differentiated cells and no cell divisions are observed.

Micronucleated cell (cmn): characterized by the presence of a main nucleus and one or more small nuclear structures called micronuclei. A micronucleus is round or almond shaped and measures between 1/3 and 1/16 of the main nucleus, has the same intensity in focal plane as the nucleus and is a fragment or a complete chromosome that at the time of mitosis is not integrated into the nucleus. one of the nuclei of the daughter cells.

Binucleate cell (bn): are cells that contain two main nuclei, usually the nuclei are very close and could even make contact, both with morphology and staining similar to a normal nucleus and there could be two cells with double genetic material.

There are few studies that include the micronucleus technique as a tool to evaluate cellular cytotoxicity in patients with metabolic syndrome or diabetes mellitus. In 2011, Andreassi et al. Studied the frequency of micronuclei in patients with obesity, diabetes and cardiovascular disease, finding greater genetic damage assessed by comet assay and micronuclei, to the group of diabetic patients and those with cardiovascular damage compared to healthy subjects ( p <0.0001 in micronucleated binuclear cells) and longer tails in patients with diabetes with cardiovascular damage compared to clinically healthy controls (p = 0.01).

In 2015, a study was conducted by Harishankar et al., Where they evaluated patients with diabetes mellitus treated with metformin and glimepiride by means of the micronucleus test in exfoliated urothelial cells, finding that those patients treated with metformin and glimepirin obtained a higher quantity of micronuclei. In comparison with healthy controls (p = 0.001) and those treated with only metformin and metformin with glimepirine, were the groups of subjects with the most micronuclei obtained, it is important to mention that they used two methods with clear field and with fluorescence stained with iodide of propidium not finding differences between both study techniques (Harishankar, 2015).

Karaman et al., In 2015, studied cytotoxic damage by comet and micronucleus assays, finding that patients with metabolic syndrome had longer tails in the comet assay (p <0.001) and also a higher number of micronuclei (p <0.001) in this same group compared to the control group.

So it would be very important to evaluate if the amount of micronuclei decreases when the patient performs a diet rich in antioxidants, because it is not yet identified if this could not only help the decrease of clinical parameters such as lipid profile, glycemic, BMI , among others; but to identify if cytotoxicity also decreases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Metabolic Syndrome that meets at least one of the ATP-III criteria:
* Abdominal obesity over 102cm for men and over 88cm for women
* Triglycerides levels over 150mg/dl with or without treatment for dyslipidemia
* c-HDL concentration under 40mg/dl for men and under 50mg/dl for women
* Blood Pressure over 130/85mmHg
* Fasting glucose levels over 100mg/dl with or without treatment

Exclusion Criteria:

* Pregnant women
* Subject with other degenerative chronic diseases does not include or consider it in ATP-III criteria for Metabolic Syndrome

Elimination Criteria

* Subjects without oral mucosa samples
* Subjects without A1c data
* Subjects without addiction to treatment under 80% with quinoa, flaxseed or both and conventional diet

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the number of micronuceli after 24 weeks | 24 weeks
  The number of micronuclei will be evaluated at baseline at 12 weeks and 24 weeks with Schmidt technique by Giemsa/wright and the entered values reflect the number of micronuclei at week 24
Changes in fasting glucose levels after 24 weeks of intervention with an added diet with quinoa or flaxseed or both or conventional diet | 24 weeks
  The fasting glucose levels will be evaluated at baseline, at 12 weeks and 24 weeks with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at 24 weeks
Changes in glycosylated hemoglobin (A1C) after 24 weeks of intervention with an added diet with quinoa or flaxseed or both or conventional diet | 24 weeks
  Glycosylated hemoglobin will be evaluated at baseline, at 12 weeks and 24 weeks by high-pressure liquid chromatography (HPLC) and the entered values reflect the glycosylated hemoglobin at 24 weeks

SECONDARY OUTCOMES:
Body Weight | 24 weeks
  The body weight will be measured at baseline, at 12 weeks and 24 weeks with a bioimpedance balance and the entered values reflect the body weight at 24 weeks
Body Mass Index | 24 weeks
  Body Mass Index will be calculated at baseline, 12 weeks and 24 weeks with the Quetelet index formula and the entered values reflect the body mass index at 24 weeks
Waist Circumference | 24 weeks
  Waist circumference will be evaluated at baseline and at 24 weeks with a flexible tape
Total Cholesterol | 24 weeks
  Total cholesterol levels will be evaluated at baseline and 24 weeks by enzymatic/colorimetric techniques and the entered values reflect the total cholesterol level at 24 weeks
Triglycerides levels | 24 weeks
  Triglycerides levels will be evaluated at baseline and 24 weeks with enzymatic/colorimetric techniques and the entered values reflect the triglycerides level at 24 weeks
High Density Lipoprotein | 24 weeks
  c-HDL levels will be evaluated at baseline and 24 weeks with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at 24 weeks
Low Density Lipoproteins | 24 weeks
  c-LDL levels will be evaluated at baseline and 24 weeks with enzymatic/colorimetric techniques and the entered values reflect the c-LDL level at 24 weeks
Blood pressure | 24 weeks
  Blood pressure will be measured at baseline and 24 weeks with a digital sphygmomanometer and the entered values reflect the blood pressure at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lilia Fletes Rayas, PhD, Principal Investigator — University of Guadalajara
Locations (2):
- Mexico (2):
  - Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco
  - Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: No
El uso de los datos es exclusivo de los investigadores involucrados en el estudio sin la devulgacion de los mismos a terceros externos al equipo de trabajo

REFERENCES:
- [Background] Andreassi MG, Barale R, Iozzo P, Picano E. The association of micronucleus frequency with obesity, diabetes and cardiovascular disease. Mutagenesis. 2011 Jan;26(1):77-83. doi: 10.1093/mutage/geq077. PMID 21164186
- [Background] Berti C, Riso P, Monti LD, Porrini M. In vitro starch digestibility and in vivo glucose response of gluten-free foods and their gluten counterparts. Eur J Nutr. 2004 Aug;43(4):198-204. doi: 10.1007/s00394-004-0459-1. Epub 2004 Jan 6. PMID 15309439
- [Background] Graf BL, Poulev A, Kuhn P, Grace MH, Lila MA, Raskin I. Quinoa seeds leach phytoecdysteroids and other compounds with anti-diabetic properties. Food Chem. 2014 Nov 15;163:178-85. doi: 10.1016/j.foodchem.2014.04.088. Epub 2014 May 4. PMID 24912714
- [Background] Ezzati M, Riboli E. Behavioral and dietary risk factors for noncommunicable diseases. N Engl J Med. 2013 Sep 5;369(10):954-64. doi: 10.1056/NEJMra1203528. No abstract available. PMID 24004122
- [Background] Karaman A, Aydin H, Geckinli B, Cetinkaya A, Karaman S. DNA damage is increased in lymphocytes of patients with metabolic syndrome. Mutat Res Genet Toxicol Environ Mutagen. 2015 Apr;782:30-5. doi: 10.1016/j.mrgentox.2015.03.009. Epub 2015 Mar 13. PMID 25868129
- [Background] Leon-Munoz LM, Guallar-Castillon P, Lopez Garcia E, Banegas JR, Gutierrez-Fisac JL, Rodriguez-Artalejo F. Relationship of BMI, waist circumference, and weight change with use of health services by older adults. Obes Res. 2005 Aug;13(8):1398-404. doi: 10.1038/oby.2005.169. PMID 16129722
- [Background] Penarrieta JM, Alvarado JA, Akesson B, Bergenstahl B. Total antioxidant capacity and content of flavonoids and other phenolic compounds in canihua (Chenopodium pallidicaule): an Andean pseudocereal. Mol Nutr Food Res. 2008 Jun;52(6):708-17. doi: 10.1002/mnfr.200700189. PMID 18537130
- [Background] Rajesha J, Murthy KN, Kumar MK, Madhusudhan B, Ravishankar GA. Antioxidant potentials of flaxseed by in vivo model. J Agric Food Chem. 2006 May 31;54(11):3794-9. doi: 10.1021/jf053048a. PMID 16719498
- [Background] Ranilla LG, Apostolidis E, Genovese MI, Lajolo FM, Shetty K. Evaluation of indigenous grains from the Peruvian Andean region for antidiabetes and antihypertension potential using in vitro methods. J Med Food. 2009 Aug;12(4):704-13. doi: 10.1089/jmf.2008.0122. PMID 19735168
- [Background] Stewart LK, Soileau JL, Ribnicky D, Wang ZQ, Raskin I, Poulev A, Majewski M, Cefalu WT, Gettys TW. Quercetin transiently increases energy expenditure but persistently decreases circulating markers of inflammation in C57BL/6J mice fed a high-fat diet. Metabolism. 2008 Jul;57(7 Suppl 1):S39-46. doi: 10.1016/j.metabol.2008.03.003. PMID 18555853
- [Background] Voss S, Hesse A, Zimmermann DJ, Sauerbruch T, von Unruh GE. Intestinal oxalate absorption is higher in idiopathic calcium oxalate stone formers than in healthy controls: measurements with the [(13)C2]oxalate absorption test. J Urol. 2006 May;175(5):1711-5. doi: 10.1016/S0022-5347(05)01001-3. PMID 16600737
- [Background] Hou Y, Aboukhatwa MA, Lei DL, Manaye K, Khan I, Luo Y. Anti-depressant natural flavonols modulate BDNF and beta amyloid in neurons and hippocampus of double TgAD mice. Neuropharmacology. 2010 May;58(6):911-20. doi: 10.1016/j.neuropharm.2009.11.002. Epub 2009 Nov 14. PMID 19917299
- See also: Epidemiología y determinantes sociales asociados a la obesidad y la diabetes tipo 2 en México — http://www.imbiomed.com.mx/1/1/articulos.php?method=showDetail&id_articulo=103591&id_seccion=329&id_ejemplar=10062&id_revista=29
- See also: NORMA Oficial Mexicana NOM-037-SSA2-2012, Para la prevención, tratamiento y control de las dislipidemias. — http://www.dof.gob.mx/nota_detalle.php?codigo=5259329&fecha=13/07/2012
- See also: Diferencias entre la prevalencia de obesidad y exceso de peso estimadas con datos declarados o por medición directa en adultos de la Comunidad Valenciana — http://scielo.isciii.es/scielo.php?script=sci_arttext&pid=S0212-16112017000100020
- See also: Nutraceuticals and Functional Foods in Health Promotion and Disease Risk Reduction — https://www.researchgate.net/publication/268288831_Nutraceuticals_and_Functional_Foods_in_Health_Promotion_and_Disease_Risk_Reduction
- See also: Utilidad de la Prueba de Micronúcleos y Anormalidades Nucleares en Células Exfoliadas de Mucosa Oral en la Evaluación de Daño Genotóxico y Citotóxico — https://scielo.conicyt.cl/scielo.php?script=sci_arttext&pid=S0717-95022013000200050
- See also: Procedimientos básicos de la prueba de micronúcleos y anormalidades nucleares en células exfoliadas de mucosa oral — http://www.medigraphic.com/cgi-bin/new/resumen.cgi?IDARTICULO=41887
- See also: Una nueva definición mundial del síndrome metabólico propuesta por la Federación Internacional de Diabetes: fundamento y resultados — http://www.revespcardiol.org/es/una-nueva-definicion-mundial-del/articulo/13082533/